CLINICAL TRIAL: NCT05920889
Title: Glucagon-like Peptide 1 Receptor Agonist in Acute Large Vessel Occlusion Stroke Treated by Reperfusion Therapies - a Pilot Study
Brief Title: Glucagon-like Peptide 1 Receptor Agonist in Acute Large Vessel Occlusion Stroke Treated by Reperfusion Therapies
Acronym: GALLOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Linyi People's Hospital (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2023.026-T
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Brain Diseases
MeSH Terms: conditions — Stroke; Ischemic Stroke; Brain Diseases | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: 140 patients will be randomized to "treatment arm" with semaglutide and standard medical therapy, and "control arm" with standard medical therapy alone in a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide Group (Active Comparator): Prescribe study drug: Patients randomized into the semaglutide group will receive 0.5mg subcutaneous injection of the drug before or during EVT, and 7 days after the procedure. i.e. semaglutide group will receive a total of 2 injections.
  Interventions: Drug: Semaglutide
- Standard of care (No Intervention): Standard medical therapy

INTERVENTIONS:
Drug: Semaglutide — 0.5mg subcutaneous injection of the drug before or during EVT, and 7 days after the procedure. i.e. patient will receive a total of 2 injections.
  Arms: Semaglutide Group

SUMMARY:
Endovascular thrombectomy (EVT) is a highly effective therapy for acute ischemic stroke with large vessel occlusion (LVO). EVT was proven efficacious in selected patients with symptoms onset or last-known-well time of up to 24 hours. With a number-needed-to-treat (NNT) of 2.3-2.8 to achieve functional independence, EVT had become the current state-of-the-art treatment for ischemic stroke with LVO. Nevertheless, more than half of LVO strokes suffered from functional dependence or death despite EVT. Futile EVTs were contributed by peri-procedural malignant brain edema (MBE) and symptomatic intracranial hemorrhage (sICH). Studies suggested that 26.9% of EVTs were complicated by MBE, whereas sICH was present in 6-9% of LVO patients who received EVT. The fundamental pathophysiology of MBE and sICH is blood-brain-barrier (BBB) disruption secondary to ischemia, mechanical and reperfusion injury. These pathological processes can result in increased tissue permeability, excess production of oxygen free radicals and inflammatory response that eventually lead to hemorrhage and edema. Poor collateral circulation, proximal LVOs, intravenous thrombolysis, blood pressure and glucose fluctuation had all been implicated to in MBE and sICH. However, these risk factors were either unmodifiable or not shown to improve EVT outcomes. The preliminary results of a recent randomized trial even suggested harmful effects of intensive blood pressure following EVT. With indications of EVT are expanding to patients with prolonged ischemia and large ischemic cores, enhancing BBB and neuronal tolerance to ischemia and reperfusion therapies may hugely impact on EVT outcomes. Recent animal models have shown that glucagon-like peptide peptide-1 receptor agonists (GLP-1RA) significantly reduced infarct volume and neurological deficits following temporary or permanent middle cerebral artery occlusion. These effects were likely due to the anti-oxidant, anti-inflammatory and anti-apoptotic properties of GLP-1RA that protected BBB integrity and ischemic neurons during induced LVO and/or reperfusion. Investigator hypothesizes that compared to standard reperfusion strategies, administration of GLP-1RA in LVO patients who receive EVT may prevent the development of MBE and sICH, and improve neurological outcomes. In this randomized, open-label pilot study, investigator aims to determine the effect of semaglutide, a GLP-1RA, on the radiological and clinical outcomes in LVO patients undergoing EVT.

DETAILED DESCRIPTION:
In this multicenter, randomized, open-label pilot study, investigator aims to recruit 140 patients with LVO strokes in the terminal internal carotid artery (ICA) or proximal middle cerebral artery (MCA) who were eligible for EVT with a last-known-well (LKW) to puncture ≤ 12 hours. Patients will be randomized in a 1:1 ratio to semaglutide or standard therapy. Patients in the semaglutide group will receive the medication on the day of (D0) and 1 week (D7) after EVT. Interval imaging and blood tests will be arranged to ascertain the degree of BBB leakage, final infarct size, inflammation and gene expression pre and post treatment. Investigator shall recruit 40 patients from the Prince of Wales Hospital and 100 patients from Linyi People's Hospital.

Detailed study procedures are as follows:-

1. LVO stroke patients will have received CTA and perfusion prior to screening.
2. Informed consent from patient or next of kin will be obtained for eligible patients.
3. After informed consent, patient will be randomized into semaglutide or standard treatment in a 1:1 ratio by computer-generated codes.
4. Patients randomized into the semaglutide group will receive 0.5mg subcutaneous injection of the drug before or during EVT, and 7 days after the procedure. i.e. semaglutide group will receive a total of 2 injections.
5. All study subjects will receive plain CT brain and perfusion D4-7 post EVT to look for MBE, sICH and hyperperfusion. Additional brain imaging may also be arranged as per clinical needs.
6. All study subjects will receive a standardized stroke protocol MRI D14-21 after EVT for quantification of infarct volume.
7. NIHSS before and immediately after, D3, D14-21, D90±7 post-EVT will be assessed.
8. mRS before, D14-21, D90±7 post-EVT will be assessed.
9. Blood test before and immediately, 3 days and 14 days after EVT (D0pre, D0post, D3, D14-21) will be collected for neurovascular inflammatory markers and transcriptomic analysis.
10. Capillary blood glucose, blood pressure and pulse will be measured four times daily in accordance to the standardized post-EVT protocol during the first 5 days hospitalization. The frequency of monitoring may increase according to the clinical needs.
11. The following data will be collected:

    1. Demographic data: date of birth, date of death (if applicable), smoking and drinking status
    2. Medical comorbidities: Hypertension, diabetes mellitus, hyperlipidemia, congestive heart failure, atrial fibrillation, ischemic heart disease, history of ischemic or hemorrhagic stroke, etc.
    3. Co-medications: Anticoagulants (apixaban, dabigatran, edoxaban, rivaroxaban, heparin, warfarin), antiplatelet agents (aspirin, clopidogrel, ticagrelor, cilostazol), lipid-lowering agents (simvastatin, atorvastatin, rosuvastatin, pravastatin, fluvastatin, ezetimibe, gemfibrozil, fenofibrate, erenumab), antihypertensive (angiotensin converting enzyme inhibitors, angiotensin receptor blockers, beta blockers, calcium channel blockers, diuretics, aldosterone antagonists, nitrates, etc.), non-steroidal antiinflammatory agents or cyclo-oxygenase2 inhibitors (indomethacin, ibuprofen, diclofenac, celecoxib, etorixocib), glucose lowering drugs (metformin, gliclazide, glimepiride, empagliflozin, dapagliflozin, insulin).
    4. Routine blood tests including hemoglobin, white cell count, lymphocyte count, neutrophil count, creatinine, alanine transferase, alkaline phosphatase, bilirubin, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, total cholesterol, triglyceride, fasting glucose, glycated hemoglobin A1c, etc. These blood tests are part of routine clinical care pre- and post-stroke.
    5. Imaging data: ASPECT score, site of occlusion, collateral score, volume of infarct core, penumbra, mismatch volume and mismatch ratio.
    6. Stroke time metrics: LKW-to-hospital, -imaging, -needle, -puncture, -reperfusion time.
    7. EVT outcomes: modified thrombolysis in cerebral infarction (TICI) score.
    8. Occurrence of MBE, asymptomatic or symptomatic ICH, hemorrhagic transformation, subarachnoid hemorrhage (see Endpoint measurement for details).

ELIGIBILITY:
Inclusion Criteria:

* LVO stroke at terminal ICA or proximal M1 eligible for emergency endovascular treatment as per current treatment guideline.
* LKW-to-puncture time ≤ 12 hours.
* Age 18 years or greater.
* National Institute of Health Stroke Scale (NIHSS) ≥10
* LVO stroke due to thromboembolism or intracranial stenosis (acute or acute on chronic occlusion).
* Patients who received computer tomographic angiography and perfusion (CTA+P).
* Pre-stroke (24 hours prior to stroke onset) independent functional status with modified Rankin Scale (mRS) ≤ 2.
* Consent process completed as per national laws and regulation and the applicable ethics committee requirements.

Exclusion Criteria:

* ASPECT score ≤ 5.
* Intracranial hemorrhage on pre-EVT imaging.
* LVO etiologies other than thromboembolism or intracranial stenosis (acute or acute on chronic total occlusion), e.g. arterial dissection, infective endocarditis on initial diagnostic imaging.Estimated or known body mass index < 18 kg/m2
* Estimated or known body mass index < 18 kg/m2.
* Pregnancy/Lactation; female, with positive urine or serum beta human chorionic gonadotropin (β-hCG) test, or breastfeeding.
* Creatinine clearance < 30mL/min.
* Severe or fatal comorbid illness, e.g. terminal malignancy.
* Participation in another clinical trial investigating a drug, medical device, or a medical procedure in the 30 days preceding trial inclusion.
* History of allergy to GLP-1RA.
* Family or personal history of multiple endocrine neoplasia, medullary thyroid carcinoma, pancreatic carcinoma, known proliferative diabetic retinopathy.
* Active sepsis on randomization.
* Patients with hypoglycaemia on presentation. Defined as capillary or serum glucose level of <4mmol/L.
* Patients prone to severe hypoglycaemia, including chronic kidney disease of estimated glomerular filtration rate of 50ml/min/1.73m^2; also those with chronic liver disease with Child's Pugh score C or above; patients with recurrent unexplained hypoglycemia.
* Patient already on GLP-1RA prior to screening.
* Contraindications to iodine-based CT contrast.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Change of Modified Rankin Score | Day 90
  Change of Modified Rankin Score to measure degree of disability/dependence. Scores 0-2 is considered good outcome, while scores 3-6 is considered poor outcome.
Composite Safety Outcome | Day 90
  Composite of Death, Intracranial Hemorrhage (ICH) and Malignant Brain Edema (MBE)

SECONDARY OUTCOMES:
Malignant brain edema (MBE) | From Day 0 post treatment, up to 90 Days.
  Parenchymal hypodensity of at least 50% of the MCA territory and signs of local brain swelling such as sulcal effacement and compression of the lateral ventricle, and Midline shift of ≥5 mm at the septum pellucidum or pineal gland with obliteration of the basal cisterns.
Symptomatic intracranial hemorrhage (sICH) | From Day 0 post treatment, up to 90 Days.
  Any parenchymal hemorrhage or hemorrhagic transformation temporally related to any worsening in neurological condition.
Blood-brain-barrier (BBB) permeability | From Day 0 post treatment, up to 90 Days.
  Blood-brain-barrier permeability by CT perfusion scan
Hemorrhagic transformation and parenchymal hemorrhage | From Day 0 post treatment, up to 90 Days.
  Hemorrhagic transformation and parenchymal hemorrhage as per Heidelberg Bleeding Classification,
Modified Rankin Score (mRS) 0-3 | From Day 0 post treatment, up to 90 Days.
  Modified Rankin Score 0-3 at 90 days
Modified Rankin Score (mRS) 0-1 | From Day 0 post treatment, up to 90 Days.
  Modified Rankin Score 0-1 at 90 days
Infarct size | Day 14-21
  Infarct size (mL) defined by brain magnetic resonance imaging segmentation
Death | Day 90
  Mortality at 90 days
Ordinal shift in Modified Rankin Score (mRS) | Day 90
  Shift in mRS at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Yiu Ming IP, MB ChB, Principal Investigator — Chinese University of Hong Kong; Fengyuan CHE, MD,PhD, Principal Investigator — Linyi People's Hospital, Shandong First Medical University & Shandong Academy of Medical Sciences
Locations (2):
- Linyi People's Hospital, Linyi, Shangdong, China
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang H, Ko H, Leung TW, Huang J, Sai J, Liang Y, Li H, Zhang J, Cao Q, Zang W, Li Y, Ma SH, Lui WT, Choi J, Chan C, Wong J, Kwok AJ, Ma K, Fan F, Chan A, Ip V, Leung H, Soo Y, Wong KT, Lai B, Chu CM, Leung HS, Hui A, Cheung T, Abrigo J, Li SH, Chan L, Yeung J, Pan S, Yip T, Lui LT, Hung T, Tsang SF, Leng X, Lam B, Mok VCT, Chan RHM, Nguyen TN, Hu W, Che F, Ip BY. Glucagon-like peptide-1 receptor agonist in large vessel occlusion treated by reperfusion therapy-a phase 2 randomized trial. Nat Commun. 2025 Dec 14;16(1):11274. doi: 10.1038/s41467-025-66167-z. PMID 41392086